CLINICAL TRIAL: NCT07330245
Title: DAHLIA: Achievement of Low Level of Disease Activity With a Dose of Corticosteroids Less Than or Equal to 5 mg (LLDAS5): a Real-life Study With Anifrolumab on Patients With Systemic Lupus Erythematosus in Italy
Brief Title: Achievement of LLDAS5 in Patients With Systemic Lupus Erythematosus Treated With Anifrolumab.
Acronym: DAHLIA
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00093
Record Dates: First submitted 2025-12-19; First posted 2026-01-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Lupus Erythematosus, Systemic.; Anifrolumab.
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Anifrolumab — anifrolumab - fully human monoclonal antibody target type I INF
  Other Names: Saphnelo

SUMMARY:
This is an observational, multicenter, prospective study on patients with systemic lupus erythematosus treated with anifrolumab in Italy aimed at evaluating the achievement of LLDAS5

DETAILED DESCRIPTION:
DAHLIA study aims to expand real-world evidence on anifrolumab role in clinical practice, specifically evaluating its effectiveness in achieving and maintenance of LLDAS with a dose of corticosteroids less than or equal to 5 mg/day (LLDAS5). Moreover it will provide data on corticosteroid tapering strategies. Additionally, will be also evaluated the Definitions Of Remission In SLE (DORIS) remission during the study period, as well as the depressive symptoms of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent to participate in the study;
* Aged 18 years or older;
* Fulfilled the 2019 EULAR/ACR classification criteria for SLE at the time of study entry;
* Prescribed anifrolumab for SLE treatment for the first time, according to the approved Italian label and reimbursement criteria;

Exclusion Criteria:

* Patients who are at LLDAS5 at the time of study entry;
* Previous exposure to anifrolumab;
* Documented diagnosis of severe or rapidly progressive Class III or IV glomerulonephritis requiring induction therapy [mycophenolate mofetil (MMF)/cyclophosphamide (CYC) + high dose steroids], isolated Class V lupus nephritis, or active severe or unstable neuropsychiatric lupus
* Currently participating in any interventional clinical trial with an investigational product;
* Inability to understand and sign the informed consent and to fill in patient questionnaires

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with Systemic Lupus Erythematous (SLE) according to 2019 EULAR/ACR classification criteria, treated with anifrolumab as per clinical practices.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of patients achieving LLDAS5 | 52 weeks
  proportion of patients with LLDAS5 at 52 weeks, defined as:
  LLDAS5 is defined as follows:
  * Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) ≤ 4, with no activity in major organ systems and no haemolytic anaemia or gastrointestinal activity;
  * No new lupus disease activity compared with previous assessment as defined per protocol;
  * Physician's Global Assessment (PGA) ≤1;
  * Current prednisone (-equivalent) dose ≤ 5mg/day;
  * Well-tolerated standard maintenance dose of immunosuppressive drugs and biologics if any.

SECONDARY OUTCOMES:
Number and percentage of patients reaching LLDAS5 at each time point | week 24, 76 and 104
  Proportion of patients with LLDAS5, according the following definition:
  LLDAS5 is defined as follows:
  * Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) ≤ 4, with no activity in major organ systems and no haemolytic anaemia or gastrointestinal activity;
  * No new lupus disease activity compared with previous assessment as defined per protocol;
  * Physician's Global Assessment (PGA) ≤1;
  * Current prednisone (-equivalent) dose ≤ 5mg/day;
  * Well-tolerated standard maintenance dose of immunosuppressive drugs and biologics if any.
Number and percentage of patients achieving a GCS (Glucocorticosterioids) dose reduction | week 4, 12, 24, 52, 76, 104 vs baseline
  Number and percentage of patients achieving a GCS dose reduction (to ≤ 5 mg/day; to 0 mg/day) at different timepoints (T1, T2, T3, T4, T5, T6) compared to T0
Median (range) cumulative dose of GCS | from week 0 to week 24; from week 24 to week 52; from week 52 to week 76; from week 76 to week 104
  Median cumulative dose of GCS calculated at each 6 month period following T0
Mean(SD) change in tender and swollen joint count | week 4, 12, 24, 52, 76 and 104 vs week 0
  Mean change in tender and swollen joint count using Disease Activity Score 28 (DAS28) map at different timepoints compared to baseline (w0). DAS28 ranges from 0 (no-activity) to 10 (high disease activity)
mean (SD) change in Power Doppler (PD) Signal Total score | week 4, 12, 24, 52, 76 and 104 vs week 0
  Mean change in Power Doppler (PD) Signal at each time point vs baseline. PD Signal ranges from 0 (low) to 84 (high)
mean (SD) change in Synovial Hypertrophy (SH) Total score | week 4, 12, 24, 52, 76 and 104 vs week 0
  Mean change in synovial hypertrophy at each time point vs baseline. Synovial hypertrophy ranges from 0 (low) to 84 (high).
Annualize flaire rate | week 52 and week 104
  Annualized flare rate in the first and second years
Number and percentage of patients meeting the DORIS clinical remission | week 12, 24, 52, 76 and 104
  Number and percentage of patients meeting the DORIS clinical remission definition at each timepoints, according to:
  * Clinical SLEDAI-2K = 0;
  * PGA < 0.5;
  * Prednisolone ≤ 5 mg/day
Number and percentage of patients with sustained DORIS remission | week 104
  Number and percentage of patients with sustained DORIS remission, defined as remaining in remission at or greater than 12 weeks after having met the DORIS definition
Mean (SD) HDRS (Hamilton Depression Rating Scale) total score | week 12, 24, 52 and 104 vs week 0
  Change in HDRS total score at different timepoints compared to T0. HDRS ranges from 0 (no depression) to 54 (severe)
Mean (SD) PROMIS Depression Short Form 8b (Patient-Reported Outcomes Measurement Information System) total score | week 12, 24, 52 and 104 vs week 0
  Change in PROMIS Depression Short Form 8b total score at different timepoints compared to week 0 (baseline). PROMIS raw scores ranges from 8 (no depression) to 40 (severe)

CONTACTS AND LOCATIONS:
Locations (19):
- Italy (19):
  - Azienda Ospedaliero-Universitaria di Cagliari Presidio di Monserrato, Monserrato, CA
  - Azienda Ospedaliero-Universitaria di Ferrara Arcispedale Sant'Anna, Cona, Ferrara
  - IRCCS Humanitas Research Hospital, Rozzano, Milano
  - AOU Ospedali Riuniti di Ancona - Presidio Torrette, Ancona
  - Azienda Ospedaliero-Universitaria Policlinico di Bari, Bari
  - ASST Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Policlinico di Modena - AOU di Modena, Modena
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera Universitaria Policlinico "Paolo Giaccone", Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero-Universitaria Pisana Ospedale Santa Chiara, Pisa
  - Policlinico Tor Vergata, Roma
  - Policlinico Umberto I - Sapienza Università di Roma, Roma
  - Azienda Ospedaliera Ordine Mauriziano Umberto I, Torino
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI) - Ospedale di Cattinara, Trieste
  - ASU Friuli Centrale - Ospedale Santa Maria della Misericordia di Udine, Udine
  - AOUI Verona - Ospedale Borgo Roma, Verona